CLINICAL TRIAL: NCT07204366
Title: Autoantibodies Against Type I Interferon in Patients Affected With Ph-negative Myeloproliferative Neoplasms (MPN-IFN Study)
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Elisa Rumi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: MPN_IFN
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Myeloproliferative Disease; COVID - 19
MeSH Terms: conditions — Myeloproliferative Disorders; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The classic Ph-negative myeloproliferative neoplasms (MPN) are a group of clonal hematopoietic disorders caused by a dysregulated JAK/STAT signal transduction because of acquired somatic mutations of JAK2, CALR or MPL genes. Chronic inflammation may predispose to MPN development.

SARS-CoV-2 infection displays extreme interindividual clinical variability, ranging from asymptomatic infection to life-threatening coronavirus disease (COVID-19). Age is a major risk factor for severe disease. Male sex and medical comorbidities have minor impact. It was demonstrated that at least 3.5% of patients with life-threatening COVID-19 have monogenic inborn errors of TLR3- or TLR7-dependent type I interferons (IFN-I) immunity. It has also been described that at least 15% of patients with life-threatening COVID-19 have neutralizing autoantibodies (AAbs) against IFN-I, that precede SARS-CoV-2 infection.

As regard MPN, COVID-19 is associated with a mortality as high as 33%. Patients with MF had the highest mortality (48%), while patients with ET had the greatest risk of venous thromboembolism (16.7%).

In this prospective study, we want to search for AAbs against IFN-I in a cohort of MPN patients to evaluate their prevalence in the MPN population and to look for clinical correlations, including COVID-19 severity.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of PV, ET, prePMF, overt PMF or MPN-U according to 2016 WHO criteria
* Characterization of the MPN driver mutation performed at any moment before enrolment
* A peripheral blood (PB) sample collected at the enrolment visit suitable for plasma extraction and functional evaluation of anti-cytokine auto-Abs

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of patients with myeloproliferative neoplasms
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate for the prevalence of AAbs neutralizing IFN-I in a cohort of Ph-neg MPN patients. | 2 years

SECONDARY OUTCOMES:
To compare the prevalence of AAbs neutralizing IFN-I in a cohort of Ph-neg MPN patients to that estimated in the general population. | 2 years
To check for association between the presence/subtype/title of AAbs to IFN-I and both clinical and molecular features of MPN patients | 2 years
To check for association between use of specific cytoreductive therapy and the presence of AAbs to IFN-I in MPN patients | 2 years
To check for association between presence/subtype/title of AAbs to IFN-I and COVID-19 severity among MPN patients who get SARS-CoV-2 infection | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No